CLINICAL TRIAL: NCT00264667
Title: A Randomised,Double-blind, Parallel Group, Placebo-controlled, Multicentre Study to Evaluate the Safety, Tolerability and Efficacy of Oral GW677954 Capsules 2.5mg, 5mg, 10mg and 20mg a Day for 24 Weeks in Overweight Dyslipidaemic Subjects
Brief Title: Study In Patients With Dyslipidaemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADG103440
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Metabolic Syndrome X
Keywords: Dyslipidaemia
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW677954

SUMMARY:
Study in patients with dyslipidaemia.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference =102cm (men) or =88cm (women) at visit 1.
* Fasting plasma HDL C =40mg/dL (1.03mmol/L) (men) or =50mg/dL (1.29mmol/L) (women) at Screening Visit 1.
* Fasting TGs =150mg/dL (1.69mmol/L) and =800mg/dL (8.96mmol/L) at Screening Visit 1.
* Subjects whose plasma LDL C concentration does not require treatment according to the NCEP ATP III guidelines at Screening Visit 1.

Exclusion Criteria:

* History of diabetes
* History of cardiovascular disease
* Diagnosis of genetic lipid disorders
* History of muscle pain
* History of cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290
Dates: Start 2005-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in non-HDL-C based on log-transformed data at week 24.

SECONDARY OUTCOMES:
Percentage change from baseline in lipids, in Homeostasis Model Assessment-insulin sensitivity (HOMA-S), C-Reactive Protein (CRP), Fasting Plasma Glucose (FPG), body weight and waist circumference.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (39):
- Argentina (5):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, San Juan
- Australia (5):
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Meadowbrook, Queensland
  - GSK Investigational Site, Elizabeth Vale, South Australia
  - GSK Investigational Site, Keswick, South Australia
  - GSK Investigational Site, Camperdown, Victoria
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- GSK Investigational Site, San José, Costa Rica
- India (4):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Mumbai
- GSK Investigational Site, Riga, Latvia
- Mexico (4):
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Pachuca, Hidalgo
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Mexico City
- New Zealand (3):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Rotorua
- Pakistan (2):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- Romania (3):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Deva
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, S.-Petresburg
- GSK Investigational Site, Košice, Slovakia
- Spain (7):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Tarrasa, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: ADG103440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ADG103440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ADG103440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ADG103440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ADG103440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ADG103440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ADG103440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register